CLINICAL TRIAL: NCT00870467
Title: A Phase 3 Multi-Center, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study Comparing Adalimumab and Placebo in Adult Japanese Subjects With Rheumatoid Arthritis
Brief Title: A Study of Adalimumab in Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-859
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- DB Placebo (Placebo Comparator): Participants received double-blind placebo administered subcutaneously (SC) every other week (eow) for up to 26 weeks. Participants also received concomitant methotrexate 6 to 8 mg administered orally weekly.
  Interventions: Drug: Double-blind Placebo
- DB adalimumab (Experimental): Participants received double-blind adalimumab 40 mg administered subcutaneously (SC) every other week (eow) for up to 26 weeks. Participants also received concomitant methotrexate 6 to 8 mg administered orally weekly.
  Interventions: Biological: Double-blind adalimumab
- DB Adalimumab/OL Adalimumab (Experimental): Participants received double-blind adalimumab administered subcutaneously (SC) every other week (eow) for 26 weeks followed by open-label adalimumab 40 mg SC eow for up to 26 weeks. Participants also received concomitant methotrexate 6 to 8 mg administered orally weekly.
  Interventions: Biological: Double-blind adalimumab; Biological: Open-label Adalimumab
- DB Placebo/OL Adalimumab (Experimental): Participants received double-blind placebo administered subcutaneously (SC) every other week (eow) for 26 weeks followed by open-label adalimumab 40 mg SC eow for up to 26 weeks. Participants received concomitant methotrexate 6 to 8 mg administered orally weekly.
  Interventions: Drug: Double-blind Placebo; Biological: Open-label Adalimumab
- DB Adalimumab/RE OL Adalimumab (Experimental): Participants received double-blind adalimumab 40 mg administered subcutaneously (SC) every other week (eow) and then open-label adalimumab 40 mg SC eow as rescue treatment (as eligible at Week 12 or after) to complete 26 weeks, followed by open-label adalimumab 40 mg SC eow for up to 26 weeks. Participants received concomitant methotrexate 6 to 8 mg administered orally weekly.
  Interventions: Biological: Double-blind adalimumab; Biological: Open-label Adalimumab; Biological: Open-labelAdalimumabRescue
- DB Placebo/RE OL Adalimumab (Experimental): Participants received double-blind placebo administered subcutaneously (SC) every other week (eow) and then open-label adalimumab 40 mg SC eow as rescue treatment (as eligible at Week 12 or after) to complete 26 weeks, followed by open-label adalimumab 40 mg SC eow for up to 26 weeks. Participants received concomitant methotrexate 6 to 8 mg administered orally weekly.
  Interventions: Drug: Double-blind Placebo; Biological: Open-label Adalimumab; Biological: Open-labelAdalimumabRescue

INTERVENTIONS:
Biological: Double-blind adalimumab — Double-blind adalimumab 40 mg administered subcutaneously (SC) every other week (eow)
  Other Names: ABT-D2E7, adalimumab, Humira
  Arms: DB Adalimumab/OL Adalimumab; DB Adalimumab/RE OL Adalimumab; DB adalimumab
Drug: Double-blind Placebo — Double-blind adalimumab-matching placebo administered subcutaneously (SC)every other week (eow)
  Other Names: Placebo
  Arms: DB Placebo; DB Placebo/OL Adalimumab; DB Placebo/RE OL Adalimumab
Biological: Open-label Adalimumab — Open-label adalimumab 40 mg administered subcutaneously (SC) every other week (eow) after completion of the first 26 weeks in the study
  Other Names: ABT-D2E7; adalimumab; Humira
  Arms: DB Adalimumab/OL Adalimumab; DB Adalimumab/RE OL Adalimumab; DB Placebo/OL Adalimumab; DB Placebo/RE OL Adalimumab
Biological: Open-labelAdalimumabRescue — Open-label adalimumab 40 mg administered subcutaneously (SC) every other week (eow) as rescue treatment to complete the first 26 weeks in the study- dependent on participant eligibility (increase in disease activity), applies to Weeks 12 to 26
  Other Names: ABT-D2E7; adalimumab; Humira
  Arms: DB Adalimumab/RE OL Adalimumab; DB Placebo/RE OL Adalimumab

SUMMARY:
To evaluate the potential of adalimumab to inhibit radiographic progression in joint destruction compared with placebo in adult Japanese subjects with recent onset of rheumatoid arthritis.

DETAILED DESCRIPTION:
This was a Phase 3 multicenter, randomized, double-blind, parallel group, placebo-controlled study designed to evaluate the inhibition of radiographic progression by adalimumab compared with placebo in adult Japanese patients with early rheumatoid arthritis (RA) who had not been previously treated with methotrexate (MTX). Eligible participants were randomized 1:1 to receive either a subcutaneous injection of adalimumab 40 mg or matching placebo every other week (eow) during the 26-week double-blind phase. All participants also received 6 mg to 8 mg MTX weekly as basal treatment for their disease. Participants who experienced an increase in disease activity (more than 20% increase in tender joint count and swollen joint count) at Week 12, 16, or 20 compared with Baseline after having increased MTX dose to 8 mg per week for at least 4 weeks were discontinued from the double-blind phase and were eligible to receive open-label adalimumab 40 mg eow as rescue treatment. Participants who completed the 26 weeks of treatment (either double-blind study drug [adalimumab or placebo] treatment or open-label adalimumab treatment) were eligible to enter the 26-week open-label phase in which they received adalimumab 40 mg eow. Efficacy and safety assessments were performed at Baseline and at designated study visits.

ELIGIBILITY:
Inclusion Criteria

* Rheumatoid arthritis based on the American College of Rheumatology criteria
* Methotrexate or leflunomide naïve
* Disease duration less than or equal to 2 years from diagnosis

Exclusion Criteria

* History of acute inflammatory joint disease of different origin from rheumatoid arthritis, cancer, lymphoma, leukemia or lymphoproliferative disease, active TB, HIV
* Previously received anti-TNF therapy anti-IL-6 receptor antibody, CTLA4-Ig, anti-CD20 antibody, cyclophosphamide, cyclosporine, azathioprine, or tacrolimus
* Joint surgery involving joints to be assessed within 8 weeks prior to Screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Ukai, BS, Study Director — Abbott Japan Co.,Ltd
Locations (88):
- Japan (88):
  - Site Reference ID/Investigator# 46861, Anjo
  - Site Reference ID/Investigator# 46919, Aomori
  - Site Reference ID/Investigator# 46805, Chiba
  - Site Reference ID/Investigator# 46806, Chiba
  - Site Reference ID/Investigator# 46880, Chiba
  - Site Reference ID/Investigator# 46881, Chiba
  - Site Reference ID/Investigator# 46890, Fuchū
  - Site Reference ID/Investigator# 46902, Fukuoka
  - Site Reference ID/Investigator# 46903, Fukuoka
  - Site Reference ID/Investigator# 46904, Fukuoka
  - Site Reference ID/Investigator# 46856, Gifu
  - Site Reference ID/Investigator# 46944, Gunma
  - Site Reference ID/Investigator# 46893, Hiroshima
  - Site Reference ID/Investigator# 46894, Hiroshima
  - Site Reference ID/Investigator# 12161, Hokkaido
  - Site Reference ID/Investigator# 46916, Hokkaido
  - Site Reference ID/Investigator# 46918, Hokkaido
  - Site Reference ID/Investigator# 46865, Hyōgo
  - Site Reference ID/Investigator# 46871, Hyōgo
  - Site Reference ID/Investigator# 46801, Ibaraki
  - Site Reference ID/Investigator# 46925, Ibaraki
  - Site Reference ID/Investigator# 46873, Kagoshima
  - Site Reference ID/Investigator# 46874, Kagoshima
  - Site Reference ID/Investigator# 46845, Kanagawa
  - Site Reference ID/Investigator# 46899, Kanagawa
  - Site Reference ID/Investigator# 46901, Kanagawa
  - Site Reference ID/Investigator# 46851, Kanazawa
  - Site Reference ID/Investigator# 46852, Kanazawa
  - Site Reference ID/Investigator# 46802, Kawagoe
  - Site Reference ID/Investigator# 46900, Kawasaki
  - Site Reference ID/Investigator# 46875, Kirishima
  - Site Reference ID/Investigator# 46870, Kitakyushu
  - Site Reference ID/Investigator# 46872, Kumamoto
  - Site Reference ID/Investigator# 46912, Kumamoto
  - Site Reference ID/Investigator# 46864, Kyoto
  - Site Reference ID/Investigator# 46943, Maebashi
  - Site Reference ID/Investigator# 46898, Matsuyama
  - Site Reference ID/Investigator# 46915, Miyazaki
  - Site Reference ID/Investigator# 46853, Nagano
  - Site Reference ID/Investigator# 46855, Nagano
  - Site Reference ID/Investigator# 46909, Nagasaki
  - Site Reference ID/Investigator# 46910, Nagasaki
  - Site Reference ID/Investigator# 46911, Nagasaki
  - Site Reference ID/Investigator# 46858, Nagoya
  - Site Reference ID/Investigator# 46860, Nagoya
  - Site Reference ID/Investigator# 46877, Nara
  - Site Reference ID/Investigator# 46885, Nara
  - Site Reference ID/Investigator# 46848, Niigata
  - Site Reference ID/Investigator# 46906, Niigata
  - Site Reference ID/Investigator# 46800, Numakunai
  - Site Reference ID/Investigator# 46869, Okayama
  - Site Reference ID/Investigator# 46886, Okayama
  - Site Reference ID/Investigator# 46887, Okayama
  - Site Reference ID/Investigator# 46892, Okayama
  - Site Reference ID/Investigator# 46876, Okinawa
  - Site Reference ID/Investigator# 46946, Osaka
  - Site Reference ID/Investigator# 46947, Osaka
  - Site Reference ID/Investigator# 46914, Ōita
  - Site Reference ID/Investigator# 46842, Rifu
  - Site Reference ID/Investigator# 46846, Sagamihara
  - Site Reference ID/Investigator# 46803, Saitama
  - Site Reference ID/Investigator# 46804, Saitama
  - Site Reference ID/Investigator# 46878, Saitama
  - Site Reference ID/Investigator# 46879, Saitama
  - Site Reference ID/Investigator# 46917, Sapporo
  - Site Reference ID/Investigator# 46942, Shimotsuke
  - Site Reference ID/Investigator# 46854, Shizuoka
  - Site Reference ID/Investigator# 46857, Shizuoka
  - Site Reference ID/Investigator# 46859, Shizuoka
  - Site Reference ID/Investigator# 46895, Takamatsu
  - Site Reference ID/Investigator# 46843, Tokyo
  - Site Reference ID/Investigator# 46844, Tokyo
  - Site Reference ID/Investigator# 46850, Tokyo
  - Site Reference ID/Investigator# 46882, Tokyo
  - Site Reference ID/Investigator# 46883, Tokyo
  - Site Reference ID/Investigator# 46884, Tokyo
  - Site Reference ID/Investigator# 46888, Tokyo
  - Site Reference ID/Investigator# 46889, Tokyo
  - Site Reference ID/Investigator# 46891, Tokyo
  - Site Reference ID/Investigator# 46896, Tokyo
  - Site Reference ID/Investigator# 46849, Toyama
  - Site Reference ID/Investigator# 46907, Toyama
  - Site Reference ID/Investigator# 46862, Toyoake
  - Site Reference ID/Investigator# 46866, Toyohashi
  - Site Reference ID/Investigator# 46863, Tsu
  - Site Reference ID/Investigator# 46926, Tsukuba
  - Site Reference ID/Investigator# 46897, Yokohama
  - Site Reference ID/Investigator# 46905, Yokohama

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778
- [Derived] Yamanaka H, Ishiguro N, Takeuchi T, Miyasaka N, Mukai M, Matsubara T, Uchida S, Akama H, Kupper H, Arora V, Tanaka Y. Recovery of clinical but not radiographic outcomes by the delayed addition of adalimumab to methotrexate-treated Japanese patients with early rheumatoid arthritis: 52-week results of the HOPEFUL-1 trial. Rheumatology (Oxford). 2014 May;53(5):904-13. doi: 10.1093/rheumatology/ket465. Epub 2014 Jan 17. PMID 24441150

RESULTS

PARTICIPANT FLOW:
Groups:
- DB Adalimumab/RE OL Adalimumab: Participants received double-blind adalimumab 40 mg administered subcutaneously (SC) every other week (eow) and then open-label adalimumab 40 mg SC eow as rescue treatment (as eligible) to complete 26 weeks, followed by open-label adalimumab 40 mg SC eow for up to 26 weeks. Participants received concomitant methotrexate 6 to 8 mg administered orally weekly.
- DB Placebo/RE OL Adalimumab: Participants received double-blind placebo administered subcutaneously (SC every other week (eow) and then open-label adalimumab 40 mg SC eow as rescue treatment (as eligible) to complete 26 weeks, followed by open-label 40 mg SC eow for up to 26 weeks. Participants received concomitant methotrexate 6 to 8 mg administered orally weekly.
Period: Double-blind
Arm/Group | DB Adalimumab | DB Placebo | DB Adalimumab/OL Adalimumab | DB Placebo/OL Adalimumab | DB Adalimumab/RE OL Adalimumab | DB Placebo/RE OL Adalimumab
Started | 171 | 163 | 0 | 0 | 0 | 0
Completed | 155 (10 participants who completed 26 weeks received open-label adalimumab 40 mg eow as rescue therapy) | 151 (24 participants who completed 26 weeks received open-label adalimumab 40 mg eow as rescue therapy) | 0 | 0 | 0 | 0
Not Completed | 16 | 12 | 0 | 0 | 0 | 0
Period: Open-label
Arm/Group | DB Adalimumab | DB Placebo | DB Adalimumab/OL Adalimumab | DB Placebo/OL Adalimumab | DB Adalimumab/RE OL Adalimumab | DB Placebo/RE OL Adalimumab
Started | 0 | 0 | 145 | 127 | 10 | 24
Completed | 0 | 0 | 132 | 120 | 5 | 21
Not Completed | 0 | 0 | 13 | 7 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Adalimumab | DB Placebo | Total
Number analyzed (Participants) | 171 | 163 | 334
Age Continuous [Mean (Standard Deviation); unit: years] | 54.0 (13.13) | 54.0 (13.20) | 54.0 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 128 | 272
  Male | 27 | 35 | 62
Region of Enrollment [Number; unit: participants]
  Japan | 171 | 163 | 334

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Total Sharp X-Ray Score at Week 26
Description: Modified Total Sharp Score (mTSS) is a measure of joint health, used in evaluation of inhibition of radiographic progression of disease. Digitized X-rays of hands and feet were obtained then scored in a blinded manner: for erosions (0 [no damage] to 5 [complete collapse or total destruction of joint]) and for joint space narrowing (0 [no damage] to 4 [complete luxation of joint]). Scores were added, giving total mTSS (0 [normal] to 380 [maximal disease]). Large positive change in mTSS indicates disease progression; small positive/no change indicates slowing/halting of disease progression.
Time Frame: Baseline, Week 26
Population: All participants who received at least 1 dose of double-blind study drug and had at least 1 efficacy assessment during double-blind study drug treatment. Analysis performed using observed cases; no imputation technique used. Participants who switched to open-label adalimumab before Week 26 were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab | DB Placebo
Number analyzed (Participants) | 148 | 128
units on a scale | 1.5 (6.07) | 2.4 (3.20)
Statistical Analysis 1: Comparison: DB Adalimumab vs DB Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants Meeting ACR20 Response Criteria at Week 26 (ACR: American College of Rheumatology)
Description: Patients were ACR20 responders if they had: >= 20% improvement in both tender joint count (68 joints) and in swollen joint count (66 joints) plus >=20% improvement in at least 3 of the 5 remaining ACR core measures: patient's assessment of pain; patient's global assessment of disease activity; physician's global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant C-reactive protein. Patients who discontinued or switched to open-label adalimumab prior to Week 26 were considered non-responders.
Time Frame: Week 26
Population: All participants who received at least 1 dose of double-blind study drug and had at least 1 efficacy assessment during double-blind study drug treatment. Non-responder imputation (NRI) performed.
Measure: Number; unit: participants
Arm/Group | DB Adalimumab | DB Placebo
Number analyzed (Participants) | 171 | 163
participants | 129 | 92
Statistical Analysis 1: Comparison: DB Adalimumab vs DB Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Number of Participants Meeting ACR50 Response Criteria at Week 26 (ACR: American College of Rheumatology)
Description: Patients were ACR50 responders if they had: >= 50% improvement in both tender joint count (68 joints) and in swollen joint count (66 joints) plus >=50% improvement in at least 3 of the 5 remaining ACR core measures: patient's assessment of pain; patient's global assessment of disease activity; physician's global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant C-reactive protein. Patients who discontinued or switched to open-label adalimumab prior to Week 26 were considered non-responders.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | DB Adalimumab | DB Placebo
Number analyzed (Participants) | 171 | 163
participants | 110 | 63
Statistical Analysis 1: Comparison: DB Adalimumab vs DB Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Secondary Outcome: Number of Participants Meeting ACR70 Response Criteria at Week 26 (ACR: American College of Rheumatology)
Description: Patients were ACR70 responders if they had: >= 70% improvement in both tender joint count (68 joints) and in swollen joint count (66 joints) plus >=70% improvement in at least 3 of the 5 remaining ACR core measures: patient's assessment of pain; patient's global assessment of disease activity; physician's global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant C-reactive protein. Patients who discontinued or switched to open-label adalimumab prior to Week 26 were considered non-responders.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | DB Adalimumab | DB Placebo
Number analyzed (Participants) | 171 | 163
participants | 81 | 37
Statistical Analysis 1: Comparison: DB Adalimumab vs DB Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

5. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28[ESR]) at Week 26
Description: Disease Activity Score (DAS28) is a combined index used to measure disease activity in patients with rheumatoid arthritis. Calculation of the DAS28 score used the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity, and the erythrocyte sedimentation rate. DAS28(ESR) scores range from 0 (no disease activity) to 9 (maximal disease activity); decrease is indicative of improvement in disease activity.
Time Frame: Baseline, Week 26
Population: All participants who received at least 1 dose of double-blind study drug and had at least 1 efficacy assessment during double-blind study drug treatment. Last observation carried forward (LOCF) was used for missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab | DB Placebo
Number analyzed (Participants) | 171 | 163
units on a scale | -2.8 (1.63) | -1.8 (1.79)
Statistical Analysis 1: Comparison: DB Adalimumab vs DB Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants Achieving Clinical Remission, Defined by Disease Activity Score (DAS28[ESR]) <2.6, at Week 26
Description: Disease Activity Score (DAS28) is a combined index used to measure disease activity in patients with rheumatoid arthritis. Calculation of the DAS28 score used the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity, and the erythrocyte sedimentation rate. DAS28(ESR) scores range from 0 (no disease activity) to 9 (maximal disease activity); decrease is indicative of improvement in disease activity. DAS28(ESR) score <2.6 was defined as clinical remission of disease.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | DB Adalimumab | DB Placebo
Number analyzed (Participants) | 171 | 163
participants | 52 | 24
Statistical Analysis 1: Comparison: DB Adalimumab vs DB Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

7. Secondary Outcome: Number of Participants Who Reported Any Adverse Event (Serious or Non-serious) on Double-blind Study Drug Through Week 26
Description: Adverse events were collected at designated study visits for all participants who were randomized and received at least 1 dose of study drug. The number of participants who experienced any adverse event (serious or non-serious) while receiving double-blind study drug is summarized. See the Reported Adverse Event section for details.
Time Frame: Through Week 26
Population: All participants who received at least 1 dose of double-blind study drug.
Measure: Number; unit: participants
Arm/Group | DB Adalimumab | DB Placebo
Number analyzed (Participants) | 171 | 163
participants | 138 | 117

8. Secondary Outcome: Change From Baseline in Modified Total Sharp X-Ray Score at Week 52
Description: Modified Total Sharp Score (mTSS) is a measure of joint health, used in evaluation of inhibition of radiographic progression of disease. Digitized X-rays of hands and feet were obtained then scored in a blinded manner: for erosions (0 [no damage] to 5 [complete collapse or total destruction of joint]) and for joint space narrowing (0 [no damage] to 4 [complete luxation of joint]). Scores were added, giving total mTSS score (0 [normal] to 380 [maximal disease]). Large positive change in mTSS indicates diseae progression; small positive/no change indicates slowing/halting of disease progression.
Time Frame: Baseline, Week 52
Population: Participants who completed 26 weeks and received at least 1 dose of adalimumab after Week 26. Analysis performed using observed cases; no imputation technique used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab/OL Adalimumab | DB Placebo/OL Adalimumab | DB Adalimumab/RE OL Adalimumab | DB Placebo/RE OL Adalimumab
Number analyzed (Participants) | 133 | 120 | 5 | 21
units on a scale | 1.6 (6.50) | 2.1 (3.25) | 9.6 (11.76) | 6.8 (9.37)

9. Secondary Outcome: Number of Participants Meeting ACR20 Response Criteria at Week 52 (ACR: American College of Rheumatology)
Description: Patients were ACR20 responders if they had: >=20% improvement in both tender joint count (68 joints) and in swollen joint count (66 joints) plus >=20% improvement in at least 3 of the 5 remaining ACR core measures: patient's assessment of pain; patient's global assessment of disease activity; physician's global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire (HAQ); and acute phase reactant C-reactive protein.
Time Frame: Week 52
Population: Participants who completed the first 26 weeks and received at least 1 dose of adalimumab after Week 26. Analysis performed using observed cases; no imputation technique used.
Measure: Number; unit: participants
Arm/Group | DB Adalimumab/OL Adalimumab | DB Placebo/OL Adalimumab | DB Adalimumab/RE OL Adalimumab | DB Placebo/RE OL Adalimumab
Number analyzed (Participants) | 133 | 120 | 5 | 21
participants | 129 | 113 | 4 | 21

10. Secondary Outcome: Number of Participants Meeting ACR50 Response Criteria at Week 52 (ACR: American College of Rheumatology)
Description: Patients were ACR50 responders if they had: >=50% improvement in both tender joint count (68 joints) and in swollen joint count (66 joints) plus >=50% improvement in at least 3 of the 5 remaining ACR core measures: patient's assessment of pain; patient's global assessment of disease activity; physician's global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire (HAQ); and acute phase reactant C-reactive protein.
Time Frame: Week 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | DB Adalimumab/OL Adalimumab | DB Placebo/OL Adalimumab | DB Adalimumab/RE OL Adalimumab | DB Placebo/RE OL Adalimumab
Number analyzed (Participants) | 133 | 120 | 5 | 21
participants | 117 | 101 | 2 | 15

11. Secondary Outcome: Number of Participants Meeting ACR70 Response Criteria at Week 52 (ACR: American College of Rheumatology)
Description: Patients were ACR70 responders if they had: >=70% improvement in both tender joint count (68 joints) and in swollen joint count (66 joints) plus >=70% improvement in at least 3 of the 5 remaining ACR core measures: patient's assessment of pain; patient's global assessment of disease activity; physician's global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire (HAQ); and acute phase reactant C-reactive protein.
Time Frame: Week 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | DB Adalimumab/OL Adalimumab | DB Placebo/OL Adalimumab | DB Adalimumab/RE OL Adalimumab | DB Placebo/RE OL Adalimumab
Number analyzed (Participants) | 133 | 120 | 5 | 21
participants | 87 | 85 | 0 | 10

12. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28[ESR]) at Week 52
Description: as for outcome 5
Time Frame: Baseline, Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab/OL Adalimumab | DB Placebo/OL Adalimumab | DB Adalimumab/RE OL Adalimumab | DB Placebo/RE OL Adalimumab
Number analyzed (Participants) | 133 | 120 | 5 | 21
units on a scale | -3.7 (1.14) | -3.7 (1.58) | -1.9 (1.22) | -3.4 (1.29)

13. Secondary Outcome: Number of Participants Achieving Clinical Remission, Defined by Disease Activity Score (DAS28[ESR]) <2.6, at Week 52
Description: as for outcome 6
Time Frame: Week 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | DB Adalimumab/OL Adalimumab | DB Placebo/OL Adalimumab | DB Adalimumab/RE OL Adalimumab | DB Placebo/RE OL Adalimumab
Number analyzed (Participants) | 133 | 120 | 5 | 21
participants | 62 | 55 | 0 | 4

14. Secondary Outcome: Number of Participants Who Reported Any Adverse Event (Serious or Non-serious) While Receiving Adalimumab Through Week 52
Description: Adverse events were collected at designated study visits for all participants who were randomized and received at least 1 dose of adalimumab. The number of participants who experienced any adverse event (serious or non-serious) while receiving any adalimumab during the study (double-blind adalimumab and/or open-label) is summarized. See the Reported Adverse Event section for details.
Time Frame: Through Week 52
Population: Participants who received at least 1 dose of adalimumab during the study.
Measure: Number; unit: participants
Groups:
- Any Adalimumab: Participants received double-blind adalimumab 40 mg administered subcutaneously (SC) every other week (eow) and/or open-label adalimumab 40 mg SC eow, including as rescue treatment.
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 326
participants | 289

ADVERSE EVENTS:
Time Frame: Through Week 26 for all participants who received at least 1 dose of blinded study drug (adalimumab or placebo) or through Week 52 for participants who received any adalimumab (double-blind and/or open-label, including rescue) in addition to methotrexate.
Description: Treatment-emergent adverse events were defined as occurring: 1) through Week 26 for Week 26 completers in blinded phase (or up to 70 days post-last dose for 26-week non-completers who never received any open-label adalimumab, including as rescue) and 2) through Week 52 for those receiving any adalimumab up to 70 days after the last adalimumab dose.
Arm/Group | DB Adalimumab | DB Placebo | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 7/171 | 4/163 | 21/326
Other Adverse Events (participants affected / at risk) | 104/171 | 83/163 | 277/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Adalimumab (N=171) | DB Placebo (N=163) | Any Adalimumab (N=326)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 4
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Facial spasm (Nervous system disorders) | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 2
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Adalimumab (N=171) | DB Placebo (N=163) | Any Adalimumab (N=326)
Constipation (Gastrointestinal disorders) | 4 | 2 | 14
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 18
Periodontitis (Gastrointestinal disorders) | 5 | 5 | 9
Stomatitis (Gastrointestinal disorders) | 6 | 15 | 17
Injection site erythema (General disorders) | 5 | 3 | 8
Injection site reaction (General disorders) | 10 | 1 | 28
Pyrexia (General disorders) | 5 | 3 | 8
Hepatic function abnormal (Hepatobiliary disorders) | 14 | 9 | 24
Liver disorder (Hepatobiliary disorders) | 4 | 3 | 9
Bronchitis (Infections and infestations) | 4 | 4 | 13
Gastroenteritis (Infections and infestations) | 2 | 4 | 8
Nasopharyngitis (Infections and infestations) | 26 | 27 | 97
Pharyngitis (Infections and infestations) | 2 | 4 | 16
Contusion (Injury, poisoning and procedural complications) | 3 | 4 | 14
Fall (Injury, poisoning and procedural complications) | 5 | 0 | 15
Alanine aminotransferase increased (Investigations) | 13 | 6 | 28
Aspartate aminotransferase increased (Investigations) | 11 | 5 | 22
Blood cholesterol increased (Investigations) | 4 | 0 | 5
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Insomnia (Psychiatric disorders) | 1 | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 28
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 4 | 7
Eczema (Skin and subcutaneous tissue disorders) | 6 | 6 | 24
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 10 | 5 | 26
Hypertension (Vascular disorders) | 5 | 8 | 12
Dental caries (Gastrointestinal disorders) | 3 | 2 | 9
Gastritis (Gastrointestinal disorders) | 2 | 1 | 10
Nausea (Gastrointestinal disorders) | 2 | 3 | 7
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 7
Cystitis (Infections and infestations) | 3 | 1 | 11
Herpes zoster (Infections and infestations) | 1 | 1 | 7
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 7
Liver function test abnormal (Investigations) | 3 | 2 | 8
White blood cell count decreased (Investigations) | 3 | 1 | 9
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 14
Dizziness (Nervous system disorders) | 1 | 3 | 7
Headache (Nervous system disorders) | 3 | 3 | 12
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.